CLINICAL TRIAL: NCT06837545
Title: Sex-specific Associations of Preoperative Serum Uric Acid Levels with Mortality and Morbidity in Non-cardiac Surgeries
Brief Title: Uric Acid and Surgical Prognosis
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ji-Hoon Sim, Assistant Professor, Asan Medical Center
Other Study IDs: AMC (2024-1090)
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Uric Acid
Keywords: Uric Acid; Mortality; Surgical Prognosis; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Other: No Intervention (Observational Study) — This study is an observational analysis of preoperative serum uric acid levels and their association with postoperative outcomes. No intervention was administered."

SUMMARY:
Preoperative serum uric acid significantly impacted mortality and morbidity in non-cardiac surgery.

DETAILED DESCRIPTION:
Preoperative SUA levels demonstrate a nonlinear, sex-specific relationship with postoperative outcomes in non-cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Patients who underwent non-cardiac surgery

Exclusion Criteria:

* Emergency surgery
* Pregnancy
* Cadavers
* Patients with missing preoperative SUA values or no follow-up after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients aged 18 years or older who underwent non-cardiac surgeries at a tertiary hospital. Patients with emergency surgeries, pregnancy, cadavers, and incomplete data with missing preoperative uric acid levels, or missing follow-up information were excluded from the analysis. The study focuses on evaluating the impact of preoperative uric acid on postoperative outcomes, including mortality and morbidities.
Sampling Method: Non-Probability Sample
Enrollment: 309353 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-02 (Actual)

PRIMARY OUTCOMES:
30-day postoperative mortality | 30 days post-surgery
  The primary outcome measure is the incidence of 30-day postoperative mortality in patients undergoing non-cardiac surgeries. Mortality is defined as death occurring within 30 days following the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa, South Korea

IPD SHARING:
Plan to Share IPD: No
The dataset used and/or analyzed during the current study is available from the corresponding author upon reasonable request.